CLINICAL TRIAL: NCT06180629
Title: The Effect Of Music During Chemotherapy On Depression, Anxiety, Stress Levels And Chemotherapy Symptoms
Brief Title: The Effect of Music During Chemotherapy
Acronym: EMDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Merve Sılgan, Nurse, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/03-08
Record Dates: First submitted 2023-11-22; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Depression; Anxiety; Stress; Chemotherapy Effect
Keywords: Depression; Stres; Anxiety; Chemotherapy Effect; Nursing; Music
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Consert (Experimental): During the chemotherapy sessions, the patients in the experimental group listened to music for 20-25 minutes, once a week for a total of 4 weeks, by choosing a music genre decided by the patient himself/herself from 3 music genres selected by the researcher based on scientific content and expert opinion.
  Interventions: Behavioral: Music conset
- control group (Active Comparator): The control group continued their normal treatment routine. No application was performed. Only pre-test and post-tests were applied.
  Interventions: Other: normal treatment routine

INTERVENTIONS:
Behavioral: Music conset — The music modes to be used (Rast and Hüseyni), classical music, nature music, and listening time of 20-30 minutes were determined by taking expert opinion from a faculty member from the Conservatory department and by reviewing the literature. The researcher asked the patients to choose the music genres. After each patient decided on the music they wanted to listen to, the researcher recorded the selected music genres on their smartphones. The music playback application was played to the patients in the experimental group for 20-25 minutes in each session for 4 sessions, i.e. 4 times in total, once a week for a month, until the end of one course. During each session, the patients listened to the music genre they had chosen each week.
  Arms: Music Consert
Other: normal treatment routine — normal treatment routine
  Arms: control group

SUMMARY:
Purpose: Chemotherapy treatment is a very different and difficult process. Considering the many physiological and psychological problems that patients experience during and after the treatment process, chemotherapy symptoms and psychological problems affect the quality of life of patients. Along with the burden of the disease, patients who experience physiological problems during chemotherapy may experience depression, stress, and anxiety. Therefore, this study was conducted to determine the effect of music played during chemotherapy on depression, anxiety, stress levels, and chemotherapy symptoms.

Method: This study was conducted in a randomized controlled manner with a pretest-posttest control group random design model. The study population consisted of patients receiving treatment in the outpatient chemotherapy unit of Maltepe University Faculty of Medicine Hospital. The study sample consisted of 49 patients who met the inclusion criteria. The power analysis determined that the sample number was 42 people in total, 21 in the experimental group and 21 in the control group. However, considering the data losses, it was decided that the number would be 25 experimental and 25 control. When one patient from the experimental group did not want to continue, the study was completed with 49 patients, 24 in the experimental group and 25 in the control group. The music recital will be applied 4 times in total, once a week, until the patients complete 1 cycle, i.e. 4 sessions. Patients in the experimental group were administered the Depression, Anxiety, Stress Scale (DASS -42) and Edmonton Symptom Diagnostic Scale (ESDS) before each session until the completion of one cycle, and music was played for 20-25 minutes during chemotherapy. After chemotherapy, the scales were applied again. In the control group, the scales were applied before chemotherapy treatment, no intervention was made during chemotherapy and the scales were applied again after chemotherapy.

DETAILED DESCRIPTION:
Population and sample: Patients who met the inclusion criteria (18 years of age or older, literate, open to communication and cooperation, having a smartphone, not having hearing problems, not in the terminal period, not receiving psychiatric treatment, receiving chemotherapy once a week, having received one course of chemotherapy, coming to the first session of the second course, and being willing and volunteering to participate in the study) were included in the study. The minimum sample size required to determine the number of patients to be assigned to the experimental and control groups was calculated using the G*Power 3.1.9.2 package program (Faul, Erdfelder, Lang et al. (2007). Considering that there may be people who may drop out of the study during the study process, it was planned to take an additional 20% sample for the study. In this case, the study sample was planned to be 50 people in total, 25 people for each of the experimental and control groups. One patient from the experimental group was excluded from the study because he did not want to continue the intervention and the study was completed with a total of 49 patients (experimental=24, control=25). Participants were numbered from 1 to 88, and 25 intervention and 25 control groups were created from the www.random.org site, taking into account the possibility of data loss.

Data collection and program application: Before starting the research, the ethics committee decision dated 02/02/2023 and numbered 2022/03-08 was taken from X Ethics Committee.

Data were collected through face-to-face interviews. Patients were asked to fill out an informed consent form before the application and their consent was obtained. Before chemotherapy started, the patients in the experimental group were informed about the music recital. Environmental factors such as light, sound and temperature were controlled and measures were taken to create a safe environment. Patient Information Form, DASS-42 Scale and ESTS were applied to the patients in both groups. After intravenous access was opened and premedication (approximately 15 minutes) was applied, they were helped to take a comfortable position in a way to maintain intravenous safety. In the experimental group, the music to be played on the patients' phones was recorded and the patient was informed. Headphones to be used for the music were provided by the researcher to the patients who did not have them. When chemotherapy started, the researcher left the patients alone during the treatment.

During the chemotherapy session; the patients in the experimental group were provided with the music of their choice during the session and the routine applications in the unit were continued, while the patients in the control group were only provided with the routine applications in the unit.

After the chemotherapy session; DASS-42 and EDSS were applied to the patients in both groups. The application continued in this way 1 time a week for a total of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Can read and write
* Open to communication and cooperation
* Having a smartphone
* No hearing problems
* Not in the terminal period
* No psychiatric treatment
* Receiving chemotherapy 1 time per week
* Patients who have received one course of chemotherapy and come to the first session of the second course
* Being willing and voluntary to participate in the research

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Depression-Anxiety-Stress Scale (DASS-42) | up to 24 weeks
  The scale consists of a total of 42 items; items with D (14 items) indicate depression, items with A (14 items) indicate anxiety, and items with S (14 items) indicate stress. The scale consists of 14 items, each answered using a 0-3 scale. Where (0) means it has never been applied to me, (3) means it has been applied to me a lot or most of the time. The normal range of scores is 0-9 for depression, 0-7 for anxiety and 0-14 for stress. Scores above these ranges indicate the degree of the problem, from mild to extreme.
Edmonton Symptom Diagnostic Scale (ESDS) | up to 24 weeks
  10 symptoms are questioned: pain, fatigue, nausea, sadness, anxiety, insomnia, loss of appetite, feeling unwell, shortness of breath and other problems. The patient is asked to match his/her symptoms with a number from 0 to 10 that he/she thinks best suits him/her. 0 indicates that he/she has no symptoms, 10 indicates that the symptom is very severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University Hospital, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No